CLINICAL TRIAL: NCT00090714
Title: To Find the Best Dose of pVGI.1(VEGF2) to Benefit Angina Patients When Given With an Experimental Injection Catheter
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Corautus Genetics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VEGF2-CAD-CL-007; NIH RAC # 0301-567
Record Dates: First submitted 2004-09-02; First posted 2004-09-06 (Estimated); Last update posted 2006-04-20 (Estimated); Status verified 2006-04

CONDITIONS: Angina Pectoris
Keywords: DNA; Circular; Gene Therapy
MeSH Terms: conditions — Angina Pectoris

INTERVENTIONS:
Genetic: pVGI.1(VEGF2)

SUMMARY:
The purpose of this study is to determine the optimum effective dose of recombinant plasmid DNA [pVGI.1(VEGF2)] gene therapy administered using an experimental cardiac direct injection catheter (Stiletto™) system needed to benefit patients with severe Angina Pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to give informed consent
* Have CCS class III or IV angina refractory to optimized medical therapy
* Experience signs or symptoms of angina during the exercise tolerance test (ETT)
* Have identified area(s) of reversible ischemic myocardium
* Have procedurally acceptable targeted treatment zones

Exclusion Criteria:

* Have exercise-limited non-cardiac chest discomfort
* Unwilling or unable to undergo exercise testing
* Able to exercise greater than 6 minutes on the treadmill
* Are candidates for conventional revascularization procedures
* Are or have been enrolled within 30 days, in another experimental study
* Have had the most recent angiogram more than 6 Months prior to screening
* Previously received an investigational angiogenic agent
* Have another disease severe enough to limit exercise test or place patient at risk
* Have uncontrolled: atrial fibrillation, atrial flutter, and/or significant arrhythmias
* Have evidence of left ventricular aneurysm or ventricular thrombus
* Are unwilling or unable to undergo cardiac catheterization or nuclear testing procedures
* Have had a Q-wave MI, within 60 days
* Have severe aortic valve stenosis or have a mechanical aortic or mitral valve
* Have unstable angina or an acute non-Q-wave myocardial infarction within 14 days
* Have had a documented stroke or transient ischemic attack within 60 days
* Are pacemaker dependent
* Have a recent history of active diabetic retinopathy or age-related wet macular degeneration
* Have a history of cancer within the last 5 yrs. or have current evidence of a malignant neoplasm
* Have a history of alcohol or drug abuse within 90 days
* Are pregnant or lactating
* Have reproductive potential and are unwilling to use condoms for contraception for 1 year after treatment - both male and female
* Are unable to return to the clinic for the scheduled follow-up appointments
* Are taking medications which may produce an undue risk
* Have areas of LV wall less than 6mm thick

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404
Dates: Start 2004-08

PRIMARY OUTCOMES:
Exercise Tolerance

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Cardiology, P.C., Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Mayo Clinic Hospital/Scottsdale, Phoenix, Arizona
  - Scripps Green Medical Center, La Jolla, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Washington Heart, Washington D.C., District of Columbia
  - Shands Hospital - Jacksonville, FL, Jacksonville, Florida
  - Crawford Long Hospital, Atlanta, Georgia
  - Fuqua Heart Center of Piedmont Hospital, Atlanta, Georgia
  - St. Joseph Hospital of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Prairie Cardiovascular, Springfield, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - Midwest CV Research Foundation, Davenport, Iowa
  - Medstar Research, Towson, Maryland
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Borgess Research Institute, Kalamazoo, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic Hospital/Rochester, Rochester, Minnesota
  - Nebraska Heart Institute, Lincoln, Nebraska
  - New York Presbyterian Hospital, New York, New York
  - Columbia Presbyterian, New York, New York
  - University of Rochester, Rochester, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Oklahoma Cardiovascular Research, Oklahoma City, Oklahoma
  - Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Baylor University Hospital, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Fletcher Allen Healthcare, Burlington, Vermont
  - Swedish Medical Center, Seattle, Washington
  - Heart Care Milwaukee, WI, Milwaukee, Wisconsin